CLINICAL TRIAL: NCT03722407
Title: A Sequential Two-Stage Dose Escalation Study to Evaluate the Safety and Efficacy of Ruxolitinib for the Treatment of Chronic Myelomonocytic Leukemia (CMML): A Phase 2 Expansion
Brief Title: Ruxolitinib for the Treatment of Chronic Myelomonocytic Leukemia (CMML): A Phase 2 Expansion
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19727
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myelomonocytic Leukemia; Leukemia
Keywords: CMML
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Leukemia | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): All patients will be given their first dose of oral Ruxolitinib, 20 mg at first scheduled visit. After that dose and on all other days patients will self-administer oral Ruxolitinib at a dose of 40 mg daily divided into two equal doses approximately 12 hours apart. Patients will be treated for a total of 16 weeks. After treatment, patients will be followed monthly.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib 5 mg tablets, 4 per dose
  Other Names: Jakafi

SUMMARY:
This study is to find out if treating Chronic Myelomonocytic Leukemia (CMML) with a study drug (ruxolitinib) can improve outcomes of patients with CMML.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Chronic Myelomonocytic Leukemia (CMML)using the World Health Organization (WHO) classification.
* 18 years of age or older at the time of obtaining informed consent.
* Must be able to adhere to the study visit schedule and other protocol requirements.
* Participants must be able to provide adequate BM aspirate and biopsy specimens for histopathological analysis and standard cytogenetic analysis during the screening procedure.
* An Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2 is required.
* Women of childbearing potential must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse 1) for at least 28 days before starting study drug; 2) while participating in the study; and 3) for at least 28 days after discontinuation from the study.
* Must understand and voluntarily sign an informed consent form.
* Must have a life expectancy of greater than 3 months at time of screening.
* Must have symptomatic splenomegaly and/or an Myeloproliferative Neoplasms Symptom Assessment Form Total Symptom Score >17.

Exclusion Criteria:

* Any of the following lab abnormalities: Platelet count of less than 35,000/uL, Absolute Neutrophil Count (ANC) less than 250/uL, Serum Creatinine ≥ 2.0, Serum total bilirubin >1.5x ULN
* Use of cytotoxic chemotherapeutic agents, or experimental agents (agents that are not commercially available) for the treatment of CMML within 28 days of the first day of study drug treatment.
* Prior history of metastatic malignancy in past 2 years
* Any serious medical condition or psychiatric illness that will prevent the subject from signing the informed consent form or will place the subject at unacceptable risk if he/she participates in the study.
* Concurrent use of Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF). Granulocyte Colony Stimulating Factor (G-CSF) could be used for the short-term management of neutropenic infection. Stable doses of erythropoietin stimulating agents that were started >8 weeks from first ruxolitinib dose or corticosteroids that were being administered prior to screening are allowed.
* Uncontrolled current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because ruxolitinib has not been studied in pregnant participants. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ruxolitinib, breastfeeding should be discontinued if the mother is treated with ruxolitinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2026-06-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Padron, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (5):
- United States (5):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Weill Medical College of Cornell University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ruxolitinib
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Response
Description: Number of participants achieving clinical benefit defined as hematologic improvement, complete remission, partial remission, or stable disease by the International Working Group Myelodysplastic/Myeloproliferative Neoplasms (MDS/MPN) Criteria.
Time Frame: At week 16
Population: Evaluable participants
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 25
Participants
  Partial Response | 3
  Marrow Response | 2
  Stable Disease | 20

2. Secondary Outcome: Time to Acute Myeloid Leukemia (AML) Transformation
Description: Time to AML transformation according to World Health Organization (WHO) Critieria
Time Frame: Every 6 months after conclusion of treatment until end of study (40.3 months)
Population: Participants who had AML transformation
Measure: Median (Full Range); unit: months
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 8
months | 5.0 [1.2 to 40.3]

3. Secondary Outcome: Overall Survival
Description: Overall survival will be from first dose of study drug until failure or death from any cause.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 29
months | 23.6 [0.2 to 24]

4. Secondary Outcome: Duration of Response
Description: Duration of response measured using time to AML transformation according to WHO Critieria
Time Frame: Up to 2 years
Population: Participants who achieved a clinical response by MDS.MPN IWG response criteria.
Measure: Median (Full Range); unit: months
Arm/Group | Ruxolitinib
Number analyzed (Participants) | 19
months | 0 [0 to 9.7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from on-study date to 30 days after end of treatment, an average of 240 days. Participants will followed for mortality for 2 years after off study date.
Arm/Group | Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 4/29
Serious Adverse Events (participants affected / at risk) | 20/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib (N=29)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Fatigue (General disorders) | 2 (2)
General disorders and administration site conditions- Other (General disorders) | 1 (1) — night sweats
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — related to COVID-19 infection
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — signs of hemoptysis
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (3) — related to COVID-19 infection
Hypoxia - related to COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat - related to COVID-19 Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Burning chest pain on exertion, related to previous COVID-19 infection
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Related to previous COVID-19 infection
Edema limbs (General disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (2)
Death, NOS (General disorders) | 4 (4)
Infections and infestations- Other (Infections and infestations) | 2 (2) — COVID-19
Gastric obstruction (Gastrointestinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ruxolitinib (N=29)
Platelet count decreased (Investigations) | 13 (43)
Aspartate aminotransferase increased (Investigations) | 11 (25)
Creatinine increased (Investigations) | 8 (26)
Alanine aminotransferase increased (Investigations) | 7 (17)
Alkaline phosphatase increased (Investigations) | 6 (18)
Neutrophil count decreased (Investigations) | 6 (19)
Blood bilirubin increased (Investigations) | 3 (7)
Investigations - Other (Investigations) | 5 (17)
White blood cell decreased (Investigations) | 3 (5)
Lymphocyte count decreased (Investigations) | 2 (5)
Cardiac troponin I increased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Edema limbs (General disorders) | 8 (8)
Fever (General disorders) | 8 (9)
Fatigue (General disorders) | 7 (7)
Pain (General disorders) | 5 (5)
Non-cardiac chest pain (General disorders) | 4 (4)
Flu like symptoms (General disorders) | 3 (6)
Chills (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (9)
Abdominal Pain (Gastrointestinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 3 (4)
Oral pain (Gastrointestinal disorders) | 3 (4)
Vomiting (Gastrointestinal disorders) | 3 (3)
Bloating (Gastrointestinal disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Obstruction gastric (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 17 (47)
Blood and lymphatic system disorders -Other (Blood and lymphatic system disorders) | 4 (10)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (16)
Metabolism and nutrition disorders -Other (Metabolism and nutrition disorders) | 4 (6)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (4)
Hyponatremia (Metabolism and nutrition disorders) | 3 (14)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (16)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 4 (4)
Infections and infestations - Other (Infections and infestations) | 3 (3)
Upper respiratory infection (Infections and infestations) | 3 (3)
Rash pustular (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3)
Bladder infection (Infections and infestations) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Gum infection (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 12 (13)
Dizziness (Nervous system disorders) | 4 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (7)
Paresthesia (Nervous system disorders) | 2 (3)
Sinus pain (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 6 (6)
Fall (Injury, poisoning and procedural complications) | 6 (7)
Fracture (Injury, poisoning and procedural complications) | 3 (3)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Intraoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 11 (16)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 5 (5)
Hot flashes (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Vascular disorders - Other (Vascular disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (4)
Urinary tract obstruction (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac disorders -Other (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Eye disorders-Other (Eye disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 (1)
Surgical and medical procedures -Other (Surgical and medical procedures) | 1 (1) — bone marrow biopsy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT03722407/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT03722407/ICF_001.pdf